CLINICAL TRIAL: NCT01151371
Title: Clinical Evaluation Of Two Daily Disposable Contact Lenses And A Monthly Replacement Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Collaborators: Visioncare Research Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-0917
Record Dates: First submitted 2010-03-24; First posted 2010-06-28 (Estimated); Results first posted 2011-12-19 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2017-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- narafilcon B daily disposable 4 weeks (Experimental): narafilcon B soft contact lenses worn daily on a daily disposable/replacement schedule, for 4 weeks
  Interventions: Device: narafilcon B contact lens
- nelfilcon A daily disponsable 1 week (Active Comparator): nelfilcon A soft contact lenses worn daily on a daily disposable/replacement schedule, for 1 week
  Interventions: Device: nelfilcon A contact lens
- lotrafilcon B daily wear, monthly replacement, 4-weeks (Active Comparator): lotrafilcon B soft contact lenses worn daily on a 1-month replacement schedule, for 4 weeks
  Interventions: Device: lotrafilcon B contact lens

INTERVENTIONS:
Device: narafilcon B contact lens — Silicone Hydrogel Daily Disposable Contact Lenses
  Arms: narafilcon B daily disposable 4 weeks
Device: nelfilcon A contact lens — Conventional Hydrogel Daily Disposable Contact Lenses
  Arms: nelfilcon A daily disponsable 1 week
Device: lotrafilcon B contact lens — Silicone Hydrogel Monthly Replacement Contact Lenses
  Arms: lotrafilcon B daily wear, monthly replacement, 4-weeks

SUMMARY:
The objective of the study is to compare the clinical performance of silicone hydrogel daily disposable contact lenses, conventional hydrogel daily disposable contact lenses and silicone hydrogel monthly replacement contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* Be no less than 18 and no more than 39 years of age.
* Sign Written Informed Consent and investigator to record this on Case Report Form (See separate document).
* Be willing and able to adhere to the instructions set out in the protocol.
* Own a cell phone and be willing to receive text messages during the day.
* Be an existing successful daily wear soft contact lens. For the purposes of this study this means wearing lenses for at least 6 hours per day, 5 days per week for the last month.
* No extended wear in the last 3 months.
* Subjective refraction must result in a vertexed spherical contact lens prescription between -1.00 and -6.00D.
* Have refractive astigmatism less than or equal to 1.00D in both eyes.
* Achieve visual acuity of 6/9 (20/30) or better in each eye.
* Require a visual correction in both eyes (no monofit or monovision allowed).
* Does not require presbyopic correction (i.e. Not using any presbyopic correction and measured add power of less than +1.00D).
* Have normal eyes with no evidence of abnormality or disease. For the purposes of this study a normal eye is defined as one having:
* No amblyopia.
* No evidence of lid abnormality or infection (including blepharitis/meibomitis).

  * No conjunctival abnormality or infection.
  * No clinically significant slit lamp findings (i.e. stromal edema, vascularization, infiltrates or abnormal opacities).
  * No other active ocular disease.

Exclusion Criteria:

* Requires concurrent ocular medication.
* Clinically significant (Grade 3 or 4) corneal stromal haze, corneal vascularization, tarsal abnormalities, bulbar hyperemia, limbal hyperemia, or any other abnormality of the cornea that would contraindicate contact lens wear.
* Clinically significant corneal staining (Grade 3 in more than one corneal region per eye).
* Requires presbyopic correction (i.e. Not using any presbyopic correction and measured add power of less than +1.00D).
* Has had refractive surgery.
* Has had eye injury/surgery within 8 weeks immediately prior to enrolment for this study.
* Abnormal lacrimal secretions.
* Pre-existing ocular irritation that would preclude contact lens fitting.
* Keratoconus or other corneal irregularity.
* PMMA(polymethyl methacrylate), hybrid or RGP(rigid gas permeable) lens wear in the previous 8 weeks.

Does not require presbyopic correction (i.e. Not using any presbyopic correction and measured add power of less than +1.00D).

* Any systemic illness which would contraindicate lens wear or the medical treatment of which would affect vision or successful lens wear.
* Diabetic.
* Infectious disease (e.g., hepatitis, tuberculosis) or an immunosuppressive disease (e.g., HIV (Human immunodeficiency virus)).
* History of chronic eye disease (e.g. glaucoma or ARMD (age related macular degeneration)).
* Pregnancy, lactating or planning a pregnancy at the time of enrolment.
* Participation in any concurrent clinical trial or in last 30 days.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 452 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2010-04-01 (Actual); Study Completion 2010-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Brea, California
  - Canoga Park, California
  - Corona, California
  - Bridgeport, Connecticut
  - Jacksonville, Florida
  - Tampa, Florida
  - Winter Park, Florida
  - Roswell, Georgia
  - Mishawaka, Indiana
  - Boston, Massachusetts
  - Blue Springs, Missouri
  - Independence, Missouri
  - Lake Ozark, Missouri
  - New York, New York
  - Raleigh, North Carolina
  - Chagrin Falls, Ohio
  - North Olmsted, Ohio
  - Warren, Ohio
  - Kittanning, Pennsylvania
  - State College, Pennsylvania
  - Warwick, Rhode Island
  - Bartlett, Tennessee
  - Brentwood, Tennessee
  - Tyler, Texas
  - Burlington, Vermont
  - Virginia Beach, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Narafilcon B 4 Weeks: lenses worn daily on a daily disposable/replacement schedule, for 4 weeks
- Nelfilcon A 1 Week: lenses worn daily on a daily disposable/replacement schedule, for 1 week
- Lotrafilcon B 4 Weeks: lenses worn daily on a 1-month replacement schedule, for 4 weeks
Period: Overall Study
Arm/Group | Narafilcon B 4 Weeks | Nelfilcon A 1 Week | Lotrafilcon B 4 Weeks
Started | 149 | 150 | 153
Completed | 144 | 149 | 146
Not Completed | 5 | 1 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Narafilcon B 4 Weeks | Nelfilcon A 1 Week | Lotrafilcon B 4 Weeks | Total
Number analyzed (Participants) | 149 | 150 | 153 | 452
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.9 (6.4) | 27.6 (6.0) | 28 (6.2) | 27.8 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 104 | 112 | 328
  Male | 37 | 46 | 41 | 124
Region of Enrollment [Number; unit: participants]
  United States | 149 | 150 | 153 | 452

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort Narafilcon B v. Nelfilcon A
Description: Contact Lens User Experience (CLUE)TM questionnaire: A validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response.
Time Frame: After 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Narafilcon B: lenses worn daily on a daily disposable/replacement schedule, for 4 weeks
- Nelfilcon A: lenses worn daily on a daily disposable/replacement schedule, for 1 week
Arm/Group | Narafilcon B | Nelfilcon A
Number analyzed (Participants) | 147 | 148
units on a scale | 68.32 (22.82) [8.4 to 21.0] | 53.75 (23.71)

2. Primary Outcome: Signs of Limbal Hyperemia Narafilcon B v. Nelfilcon A
Description: Redness scale of 0 to 4, where 0=None, 4=Severe redness
Time Frame: After 1 Week
Measure: Mean (Standard Deviation); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | Narafilcon B | Nelfilcon A
Number analyzed (Participants) | 147 | 148
Number analyzed (eyes) | 294 | 296
Units on a scale | 0.53 (0.50) | 0.61 (0.51)

3. Primary Outcome: Subjective Rating of Overall Comfort Narafilcon B v. Lotrafilcon B
Description: as for outcome 1
Time Frame: After 4 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lotrafilcon B: lenses worn daily on a 1-month replacement schedule, for 4 weeks
Arm/Group | Narafilcon B | Lotrafilcon B
Number analyzed (Participants) | 142 | 143
units on a scale | 66.43 (23.37) | 53.91 (23.72)

4. Secondary Outcome: Signs of Inferior Corneal Staining Narafilcon B v. Nelfilcon A
Description: Standard scale of 0 to 3 where 0=None, 3=Severe staining
Time Frame: After 1 Week
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Narafilcon B | Nelfilcon A
Number analyzed (Participants) | 147 | 148
Number analyzed (eyes) | 294 | 296
units on a scale | 0.13 (0.36) | 0.31 (0.57)

5. Secondary Outcome: Subjective Rating of Overall Ease of Lens Handling Narafilcon B v Nelfilcon A
Description: as for outcome 1
Time Frame: After 1 Week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Narafilcon B | Nelfilcon A
Number analyzed (Participants) | 147 | 148
units on a scale | 64.05 (22.35) | 60.76 (22.03)

6. Secondary Outcome: Subjective Rating of End of Day Comfort Narafilcon B v. Nelfilcon A
Description: Scale of 1 to 5, where 1=Poor comfort and 5=Excellent comfort
Time Frame: After 1 Week
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Narafilcon B | Nelfilcon A
Number analyzed (Participants) | 147 | 148
units on a scale | 3.69 (0.11) | 2.81 (0.11)

7. Secondary Outcome: Subjective Rating of Initial Comfort Narafilcon B v. Nelfilcon A
Description: Comfort immediately after the lens is put on the eye. Scale of 1 to 5, where 1=poor comfort and 5=excellent comfort.
Time Frame: After 1 Week
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Narafilcon B | Nelfilcon A
Number analyzed (Participants) | 147 | 148
units on a scale | 4.10 (0.13) | 3.92 (010)

8. Secondary Outcome: Signs of Inferior Corneal Staining Narafilcon B v. Lotrafilcon B
Description: Scale of 0 to 3, where 0=none and 3=severe staining.
Time Frame: After 4 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Narafilcon B | Lotrafilcon B
Number analyzed (Participants) | 147 | 148
units on a scale | 0.14 (0.41) | 0.34 (0.60)

9. Secondary Outcome: Subjective Rating of Overall Ease of Lens Handling Narafilcon B v. Lotrafilcon B
Description: as for outcome 1
Time Frame: After 4 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Narafilcon B | Lotrafilcon B
Number analyzed (Participants) | 147 | 148
units on a scale | 62.58 (22.79) | 55.50 (22.47)

10. Secondary Outcome: Subjective Rating of End of Day Comfort Narafilcon B v. Lotrafilcon B
Description: Scale of 1 to 5, where 1=poor comfort and 5=excellent comfort
Time Frame: After 4 Weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Narafilcon B | Lotrafilcon B
Number analyzed (Participants) | 147 | 148
units on a scale | 3.55 (0.11) | 2.95 (0.11)

11. Secondary Outcome: Subjective Rating of Initial Comfort Narafilcon B v. Lotrafilcon B
Description: Comfort immediately after the lens is put on the eye. Scale of 1 to 5, where 1=poor comfort, 5=excellent comfort.
Time Frame: After 4 Weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Narafilcon B | Lotrafilcon B
Number analyzed (Participants) | 147 | 148
units on a scale | 4.25 (0.10) | 3.79 (0.09)

12. Primary Outcome: Signs of Limbal Hyperemia Narafilcon B v. Lotrafilcon B
Description: Redness scale of 0 to 4, where 0=None, and 4=Severe.
Time Frame: After 4 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | Narafilcon B | Lotrafilcon B
Number analyzed (Participants) | 142 | 143
Number analyzed (eyes) | 284 | 286
units on a scale | 0.44 (0.47) | 0.68 (0.61)

ADVERSE EVENTS:
Arm/Group | Narafilcon B 4 Weeks | Nelfilcon A 1 Week | Lotrafilcon B 4 Weeks
Serious Adverse Events (participants affected / at risk) | 0/149 | 0/150 | 0/153
Other Adverse Events (participants affected / at risk) | 0/149 | 0/150 | 0/153

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must provide written approval for any publication.